CLINICAL TRIAL: NCT03161704
Title: Validation and Refinement of Noninvasive Diagnostic Biomarkers for Endometriosis, The ENDOmarker Protocol
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Augusta University (Other); Penn State University (Other); University of California, San Francisco (Other); University of North Carolina (Other); University of Oklahoma (Other); University of Pennsylvania (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ENDOmarker
Record Dates: First submitted 2015-11-13; First posted 2017-05-22 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Collection of endometrial biopsy tissue, serum, plasma, whole blood for DNA extraction and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study involves the prospective collection of endometrial biopsy tissue, serum, plasma, whole blood for DNA extraction, and urine from women who will be diagnosed as having (or not having) endometriosis at the time of scheduled surgery. The investigators plan to enroll approximately 500 women to validate and optimize the use of genomic classifiers alone or in combination with serum markers (such as cytokines) as a non-surgical marker of disease.

ELIGIBILITY:
Exclusion Criteria:

* • Currently pregnant

  * Current or past diagnosis of any malignancy (with the exception of non-melanoma skin cancer)
  * Known to be HIV-positive
  * Unable to give informed consent
  * Unwillingness to have samples banked in Repository for future use
  * Clinical evidence of active cervical infection
  * Lupron (or other GRH agonist) therapy within the last 2 months (or Depo-Lupron within the last 4 months)
  * Current use of estrogen or progestin (oral, transdermal, intrauterine or ring).

    o Current use is defined as use in the index menstrual cycle (since the onset of the last menstrual period).
  * Use of depo estrogen or progestin in last 3 months
  * Current use of aromatase inhibitor

Inclusion Criteria:

* Women aged 18-44 scheduled to undergo gynecologic surgery (laparoscopy/laparotomy).

Indication for surgery can include: infertility, endometriosis, tubal ligation, lysis of adhesions, pelvic pain, hysterectomy (for benign condition), myomectomy, salpingo-oophorectomy, cystectomy, or diagnostic laparoscopy.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females aged 18-44 who are scheduled to undergo gynecologic surgery (laparoscopy/laparotomy). Indications for surgery can include: infertility, endometriosis, tubal ligation, lysis of adhesions, pelvic pain, hysterectomy (for benign condition), myomectomy, salpingo-oophorectomy, cystectomy, or diagnostic laparoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Collection of up to 3 2cm samples of Endometrial Tissue | 2 collection timepoints: baseline and up to 18 weeks following surgery.
  Up to 3 2cm samples will be collected per collection.

SECONDARY OUTCOMES:
Collection of Serum 1 will be 2 10ml serum tubes of serum | 3 collection timepoints: baseline, up to 14 days following surgery and up to 18 weeks following surgery.
  2 10ml serum tubes will be drawn at each collection, up to 10 1.0ml aliquots per collection.
Collection of Serum 2 will be 2 7 ml serum tubes of serum | 3 collection timepoints: baseline, up to 14 days following surgery and up to 18 weeks following surgery.
  2 7ml serum tubes drawn at each collection, up to 10 1.0ml aliquots of serum plus 1 15ml conical tube with the 2 blood clots per collection.

OTHER OUTCOMES:
Collection of Plasma in 1 4ml EDTA tube | 3 collection timepoints: baseline, up to 14 days following surgery and up to 18 weeks following surgery.
  1 4ml EDTA tube will be drawn at each collection, up to 3 1.0ml aliquots per collection.
Collection of Whole Blood in 2 4ml EDTA tubes | 3 collection timepoints: baseline, up to 14 days following surgery and up to 18 weeks following surgery.
  2 4ml EDTA tubes will be drawn at each collection, up to 2 4.5ml aliquots as well as 1 FTA blood spot collection card per collection.
Collection of Urine will be one complete sample as produced by the subject | 3 collection timepoints: baseline, up to 14 days following surgery and up to 18 weeks following surgery.
  1 urine sample will be collected each time, up to 6 15ml aliquots and 5 1.5ml aliquots per collection will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Barnhart, MD MSCE, Principal Investigator — University of Pennsylvania; Esther Eisenberg, MD MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Michael Diamond, MD, Principal Investigator — Augusta University; Richard Legro, MD, Principal Investigator — Milton S. Hershey Medical Center; Marcelle Cedars, MD, Principal Investigator — University of California, San Francisco; Anne Steiner, MD MPH, Principal Investigator — University of North Carolina; Karl Hansen, MD PhD, Principal Investigator — University of Oklahoma; Christos Coutifaris, MD PhD, Principal Investigator — University of Pennsylvania; Heping Zhang, PhD, Principal Investigator — Yale University
Locations (5):
- United States (5):
  - Yale University, New Haven, Connecticut
  - Augusta University, Augusta, Georgia
  - Wayne State University, Southfield, Michigan
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania